CLINICAL TRIAL: NCT04093713
Title: Inferior Alveolar Nerve Block: a Novel Intraoral Technique Depends on Extraoral Landmarks
Brief Title: A Novel Technique to Anaesthetize the Lower Jaw
Acronym: NTALJ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mosaad Khalifah (Other)
Responsible Party: Sponsor-Investigator, Mosaad Khalifah, Lecturer and researcher, Hosh Isa Medical Center
Organization: Hosh Isa Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Surg192
Record Dates: First submitted 2019-09-13; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Inferior Alveolar Nerve Block
Keywords: Anaesthesia; Technique; extraoral; Landmarks
MeSH Terms: interventions — Nordefrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- participants (Other): participants are subjected to a novel technique to block the inferior alveolar nerve depending on extraoral landmarks
  Interventions: Procedure: A novel technique to block the inferior alveolar nerve block using Mepivecaine with Levonordefrin

INTERVENTIONS:
Procedure: A novel technique to block the inferior alveolar nerve block using Mepivecaine with Levonordefrin — blocking the inferior alveolar nerve using extroral landmarks

SUMMARY:
This study introduces and evaluates a new technique for inferior alveolar nerve blocking.

DETAILED DESCRIPTION:
The study addresses a novel technique to anaesthetize the inferior alveolar nerve depending on extraoral landmarks. Volunteers will receive bilateral blocks and evaluation of the success rate and positive aspiration rate will be performed.

ELIGIBILITY:
Inclusion Criteria:

* fitness for nerve block local anaesthesia physically and psychologically

Exclusion Criteria:

* any disease or condition obstacles nerve block local anaesthesia administration such as hemophilia.

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 65 (Estimated)
Dates: Start 2019-09-14 (Estimated); Primary Completion 2019-09-16 (Estimated); Study Completion 2019-09-16 (Estimated)

PRIMARY OUTCOMES:
presence of numbness (by questionnaire) | 3-10 minutes
  evaluation of the presence of numbness in the anatomical area supplied by the inferior alveolar nerve
absence of pain (by probing) | 3-10 minutes
  evaluation of absence of pain in the anatomical area supplied by the inferior alveolar nerve

SECONDARY OUTCOMES:
positive aspiration rate | 1 second
  evaluation of the presence of blood on drawing in two perpendicular planes

CONTACTS AND LOCATIONS:
Overall Officials: Mosaad A Khalifah, DDSc, Principal Investigator — Kafrelsheikh University
Locations (1):
- Hosh Isa Medical Center, Ḩawsh ‘Īsá, Al-Behera, Egypt

IPD SHARING:
Plan to Share IPD: No
No other researchers are involved in the study

REFERENCES:
- [Background] Kanaa MD, Whitworth JM, Corbett IP, Meechan JG. Articaine buccal infiltration enhances the effectiveness of lidocaine inferior alveolar nerve block. Int Endod J. 2009 Mar;42(3):238-46. doi: 10.1111/j.1365-2591.2008.01507.x. PMID 19228214
- [Background] Donkor P, Wong J, Punnia-Moorthy A. An evaluation of the closed mouth mandibular block technique. Int J Oral Maxillofac Surg. 1990 Aug;19(4):216-9. doi: 10.1016/s0901-5027(05)80395-9. PMID 2120362
- [Background] Montagnese TA, Reader A, Melfi R. A comparative study of the Gow-Gates technique and a standard technique for mandibular anesthesia. J Endod. 1984 Apr;10(4):158-63. doi: 10.1016/S0099-2399(84)80120-X. No abstract available. PMID 6586971
- [Background] McLean C, Reader A, Beck M, Meryers WJ. An evaluation of 4% prilocaine and 3% mepivacaine compared with 2% lidocaine (1:100,000 epinephrine) for inferior alveolar nerve block. J Endod. 1993 Mar;19(3):146-50. doi: 10.1016/s0099-2399(06)80510-8. PMID 8509754
- [Background] Akinosi JO. A new approach to the mandibular nerve block. Br J Oral Surg. 1977 Jul;15(1):83-7. doi: 10.1016/0007-117x(77)90011-7. PMID 268212
- [Background] Boonsiriseth K, Sirintawat N, Arunakul K, Wongsirichat N. Comparative study of the novel and conventional injection approach for inferior alveolar nerve block. Int J Oral Maxillofac Surg. 2013 Jul;42(7):852-6. doi: 10.1016/j.ijom.2012.11.017. Epub 2012 Dec 21. PMID 23265758
- [Background] Suazo Galdames IC, Cantin Lopez MG, Zavando Matamala DA. Inferior alveolar nerve block anesthesia via the retromolar triangle, an alternative for patients with blood dyscrasias. Med Oral Patol Oral Cir Bucal. 2008 Jan 1;13(1):E43-7. PMID 18167480